CLINICAL TRIAL: NCT06491212
Title: Examination of Diaphragm Function, Postural Control, and Plantar Pressure in Individuals With Pes Planus
Brief Title: The Relationship Between Pes Planus, Diaphragm, Postural Control, and Plantar Pressure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Ayça Araci, Assistant professor, Alanya Alaaddin Keykubat University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 8880-GOA
Record Dates: First submitted 2024-06-24; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Pes Planus; Diaphragm Issues; Plantar Pressure; Postural Control
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Intervention Model Description: Our study was planned to evaluate healthy controls and cases with pes planus.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- People with pes planus (Experimental): Individuals with pes planus that we identified according to the inclusion criteria will be evaluated in this group.
  Interventions: Diagnostic Test: Determination of Foot Deformity Level; Diagnostic Test: Foot Function Index; Diagnostic Test: UFAA-International Physical Activity Questionnaire; Diagnostic Test: Diaphragm ultrasound measurements; Diagnostic Test: NeuruCom Balance Master Balnce and Performans Test; Diagnostic Test: Plantar Pressure Assessment
- Healthy People (Active Comparator): Volunteer individuals without pes planus who meet the inclusion criteria will be evaluated for comparison in this group
  Interventions: Diagnostic Test: Determination of Foot Deformity Level; Diagnostic Test: Foot Function Index; Diagnostic Test: UFAA-International Physical Activity Questionnaire; Diagnostic Test: Diaphragm ultrasound measurements; Diagnostic Test: NeuruCom Balance Master Balnce and Performans Test; Diagnostic Test: Plantar Pressure Assessment

INTERVENTIONS:
Diagnostic Test: Determination of Foot Deformity Level — One of the methods used in our study to determine the presence and degree of pes planus is the navicular drop test.
Diagnostic Test: Foot Function Index — Evaluation of Foot Function
Diagnostic Test: UFAA-International Physical Activity Questionnaire — To determination of physical activity level.
Diagnostic Test: Diaphragm ultrasound measurements — Rehabilitative ultrasound imaging is a method frequently used by physiotherapists to assess muscle function.
Diagnostic Test: NeuruCom Balance Master Balnce and Performans Test — Balance master will be used for postural stability, static and dynamic balance measurements.
Diagnostic Test: Plantar Pressure Assessment — When assessing plantar pressure, postural control will be evaluated statically or dynamically, through examination of the behavior of the center of plantar pressure (COP).

SUMMARY:
Our primary aim is to compare diaphragm function (resting thickness, activity/resting thickness ratio indicating contractility), postural control, and plantar pressure between individuals with pes planus and healthy controls without pes planus.

DETAILED DESCRIPTION:
Pes planus deformity, by causing pronation during standing, affects the biomechanics of the lower extremities. Improper foot positioning can lead to changes in load distribution under the sole, and consequently, abnormal tensions in the soft tissues of the feet can spread to the upper body parts through the myofascial system. In light of all this information, our primary aim is to examine the diaphragm function and thickness in individuals with pes planus deformity and healthy individuals, and to investigate the relationship between diaphragm thickness and balance. Additionally, our secondary aim is to evaluate the relationship between pes planus, diaphragm thickness, and balance.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for individuals with Pes Planus Deformity

* Willing to participate in the study voluntarily
* Having a Navicular drop test value of 10mm or above
* Being between the ages of 18-30
* Having the physical capacity to perform assessments and tests
* Having a body mass index of 18-25 kg/m²

Exclusion Criteria:

* Exclusion criteria for individuals with Pes Planus Deformity:
* Termination of voluntariness
* Those with rigid flatfoot, pes cavus, hallux valgus, hallux rigidus, or calcaneal spur deformity
* Those with chronic systematic and metabolic diseases (e.g., diabetes mellitus, rheumatoid arthritis, etc.) and musculoskeletal problems (e.g., pes planus) that may affect foot functions and gait
* Those with any surgical history likely to affect balance, lower extremity strength, and postural control
* Those with any visual/vestibular, musculoskeletal, or neurological problems"

Inclusion criteria for healthy participants:

* Willing to participate in the study voluntarily
* Being between the ages of 18-30
* Having the physical capacity to perform assessments and tests
* Having a body mass index of 18-25 kg/m²
* Having the ideal height of the medial longitudinal arch of the foot (not having pes planus)

Exclusion criteria for healthy participants:

* Termination of voluntariness
* Those with chronic systematic and metabolic diseases (e.g., diabetes mellitus, rheumatoid arthritis, etc.) and musculoskeletal problems (e.g., pes planus) that may affect foot functions and gait
* Those with any surgical history likely to affect balance, lower extremity strength, and postural control
* Those with any visual/vestibular, musculoskeletal, or neurological problems"

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Navicular Drop Test | The evaluation will be conducted once and will be completed within 12 months.
  One of the methods used in our study to determine the presence and degree of pes planus is the navicular drop test. If the navicular height difference is between 6-9 mm, it is considered normal MLA, and if it is 10 mm or more, it is considered pes planus.
Foot Function Index | The evaluation will be conducted once and will be completed within 12 months.
  The Foot Function Index consists of 3 subscales: pain, disability and activity limitation. The pain subscale, consisting of nine items, measures the level of foot pain in various situations, while the disability subscale determines the degree of difficulty in performing various functional activities due to foot problems. The five-item activity limitation subscale assesses limitations in activities due to foot problems. Individuals score all items using the Visual Analog Scale (VAS), taking into account their foot condition one week ago. To calculate subscale and total scores, the score for each item is summed, divided by the sum of the maximum scores of the items and multiplied by 100. Higher scores indicate more pain, disability and activity limitation.
UFAA-International Physical Activity Questionnaire | TThe evaluation will be conducted once and will be completed within 12 months.
  In our study, the self-administered short form of the questionnaire, which includes the "last seven days", will be used to assess physical activity level. Minutes, days and METs (multiples of resting oxygen consumption) are multiplied to obtain a score as "MET-minutes/week". Physical activity levels are classified as physically inactive (<600 MET-min/week), low physical activity (600 - 3000 MET-min/week) and adequate physical activity (>3000 MET-min/week). In the calculation of energy expenditure for physical activities, the weekly duration (minutes) of each activity is multiplied by the MET energy values created for the International Physical Activity Questionnaire. Thus, energy expenditures for vigorous, moderate, walking, sitting and total physical activities for each individual are obtained in MET-min/week.
Evaluation of Diaphragmatic Functions | The evaluation will be conducted once and will be completed within 12 months.
  The evaluations will be performed with B-mode for bilateral hemidiaphragm in the supine position of the participant. Thickness measurements will be made between hyperechoic peritoneal and pleural borders and recorded in mm (24,25). The thickening fraction (%), which shows the constrictibility of the muscle, in other words, the change in thickness, will be calculated using the formula "(deep inspiration thickness-calm expiration thickness) x 100 / calm expiration thickness
Evaluation Balance | The evaluation will be conducted once and will be completed within 12 months.
  NeuroCom Balance Master balance and performance test device (NeuroCom System Version 8.1.0, B 100718, 1989- 2004 NeuroCom® International Inc. USA) will be used for the evaluation of balance. Balance master is a valid and reliable test device widely used in postural stability, static and dynamic balance measurements.
Plantar Pressure Assessment | The evaluation will be conducted once and will be completed within 12 months.
  Tekscan MatScan™ Pressure Mat System (Tekscan Inc. Boston, USA) will be used to evaluate plantar pressure in the study.The assessments will be performed statically and dynamically. COF ellipse area (cm2), COF velocity (cm/s), COF deviation length (cm), anteroposterior deviation COFx (cm), mediolateral deviation COFy (cm) data obtained in the evaluations and weight values for right-left and anteroposterior feet will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Alanyaaku, Antalya, Alanya, Turkey (Türkiye)